CLINICAL TRIAL: NCT06180187
Title: Radiographic and Clinical Comparative Study Between Osseodensification Burs and Electrical Mallet in Closed Sinus Floor Elevation and Simultaneous Implant Placement. Prospective Clinical Trial.
Brief Title: Densah Burs vs. Electrical Mallet in Closed Sinus Lifting.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Abdelrahman sayed mostafa elsayed, Dentist, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1222023
Record Dates: First submitted 2023-12-04; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Alveolar Bone Loss
Keywords: sinus lift; electrical mallet; osseodensification; bone density
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: group I (Osseo Densification group) Patients in this group will have sinus floor elevation using osseodensification burs then application of PRF membrane through the socket to protect schneiderian membrane and application of sticky bone (xeno graft and i-PRF) to augment alveolar ridge to receive dental implant
  group II (electrical mallet group) Patients in this group will have sinus floor elevation using electrical mallet then application of PRF membrane through the socket to protect schneiderian membrane and application of sticky bone (xeno graft and i-PRF) to augment alveolar ridge to receive dental implant
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osseo-densification group (Active Comparator)
  Interventions: Device: Osseo-densification burs
- Electrical mallet group (Active Comparator)
  Interventions: Device: Electrical mallet

INTERVENTIONS:
Device: Electrical mallet — elevation of the Schneiderian membrane of maxillary sinus using electrical mallet and place bone graft material to augment the residual alveolar ridge and then place dental implant .
  Arms: Electrical mallet group
Device: Osseo-densification burs — elevation of the Schneiderian membrane of maxillary sinus using osseodensification burs and place bone graft material to augment the residual alveolar ridge and then place dental implant .
  Arms: Osseo-densification group

SUMMARY:
The aim of the comparative study is to evaluate the density and amount of new bone formed (bone height gain)around dental implant placed simultaneously in posterior maxilla after closed sinus floor elevation using Osseodensification burs versus electrical mallet.

DETAILED DESCRIPTION:
Extraction of posterior teeth in the maxilla for long time without rehabilitation of the area increases the incidence of maxillary sinus pneumatization that makes maxillary sinus enlarges in volume over the residual bone of alveolar ridge.

Decreasing the height of sub_ antral bone affects adversely on the bone density which is crucial for implant primary stability causing placement of dental implant quite challenging requiring sinus lifting procedure and bone condensation of residual ridge in addition to bone grafting

Summers technique considered the gold standard for closed sinus floor elevation using osteotome and a hand mallet to condense alveolar bone and elevate schneiderian membrane. One of drawbacks of this technique is benign paroxysmal positional vertigo due to force applied by hand mallet is not controlled.

Electrical mallet was introduced to overcome (BPPV) as it applies controlled force (daN) in short fraction of seconds(µs) with hand piece secured totally by the surgeon and have a wide variety of instruments placed on the hand piece e.g. osteotomes used in sinus floor elevation .

Controlled force of magnetic mallet decrees the risk of schneiderian membrane perforation

Osseodensification burs now show great outcomes in closed sinus lifting procedure.

Densah burs increase the density of alveolar bone which increase the primary stability of dental implants .

Aim of this study is to compare Electrical mallet with Osseodensification burs in closed sinus lifting.

ELIGIBILITY:
Inclusion Criteria:

* patients with partially edentulous posterior maxilla
* Residual bone height ≥ 5mm
* Oral hygiene : fair oral hygiene

Exclusion Criteria:

* Smoking
* Systematic disease that affects bone remodeling (e.g. uncontrolled Diabetes mellitus or osteoporosis)
* Radiotherapy to head and neck or chemotherapy
* Chronic disease of maxillary sinus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
bone height gain | 6 months follow up
  Evaluate the change in bone height radiographically after closed sinus floor elevation and simultaneous implant placement .using cone beam computed tomography immediate after surgery and 6 months post operative .
change in bone density | 6 months follow up
  Evaluate the amount of change in bone density around dental implant immediately post operative and after 6 months.